CLINICAL TRIAL: NCT06042036
Title: Adherence to Low Tidal Volume in the Transition to Spontaneous Ventilation Mode in Patients With Acute Respiratory Failure in ICUs in Latin America
Brief Title: Adherence to Low Tidal Volume in the Transition to Spontaneous Ventilation in Patients With Acute Respiratory Failure
Acronym: SPIRAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Brazilian Research In Intensive Care Network (Network); Latin American Intensive Care Network (LIVEN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 28482720.0.1001.0068
Record Dates: First submitted 2023-09-04; First posted 2023-09-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-09

CONDITIONS: Respiration, Artificial; Acute Hypoxemic Respiratory Failure; Respiratory Insufficiency
Keywords: Adherence, Treatment; intensive care units
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute hypoxemic respiratory failure: Patients with acute hypoxemic respiratory failure transitioning to a spontaneous mode of mechanical ventilation ( PSV, APRV, NAVA, PAV+, CPAP)
  Interventions: Other: Spontaneous mode of mechanical ventilation

INTERVENTIONS:
Other: Spontaneous mode of mechanical ventilation — any mode of mechanical ventilation classified as spontaneous or proportional, mainly pressure support ventilation, but also CPAP, APRV, NAVA, PAV+
  Other Names: spontaneous ventilation

SUMMARY:
The goal of this observational study is to estimate the prevalence of the use of protective ventilation with low tidal volume ventilation in the transition of spontaneous ventilation modes in patients with hypoxemic acute respiratory failure in ICUs in Latin America and its association with patient outcomes.

The main questions it aims to answer are:

* what is the prevalence of the use of low tidal volume ventilation (VT <8 mL/kg of predicted body weight) in the first 24 hours of spontaneous ventilation modes in patients with hypoxemic acute respiratory failure?
* Is there an association between the rate of adherence to low tidal volume ventilation in spontaneous ventilation modes and the ability to stay off ventilatory support and mortality?

Participants are patients with acute respiratory failure under mechanical ventilation. Investigators will collect data on the ventilatory parameters of participants

* 24 hours before they begin to be ventilated with spontaneous modes of ventilation
* during the first 24 hours of spontaneous ventilation

Investigators will collect several patient-centered clinical outcomes at 28 days after study inclusion, including ventilator-free days and mortality

DETAILED DESCRIPTION:
Investigators will conduct a cohort study in Intensive Care Units (ICUs) across Latin America, aiming to include 422 patients with Hypoxemic Acute Respiratory Failure (ARF) and under invasive mechanical ventilation.

The goal of this observational study is to estimate the prevalence of the use of protective ventilation with low tidal volume ventilation in the transition of spontaneous ventilation modes in patients with hypoxemic acute respiratory failure in ICUs in Latin America

The primary objectives are to determine the prevalence of low tidal volume ventilation (VT < 8 mL/kg of predicted body weight) during the initial 24 hours of spontaneous ventilatory modes in patients diagnosed with hypoxemic ARF and its association with clinically important patient outcomes. Investigators are interested in assessing the rate of adherence to low tidal volume ventilation, defined as maintaining VT < 8 mL/kg of predicted body weight during the first 24 hours of ventilation in spontaneous mode.They are also interested in measuring the number of days that patients are alive and not receiving ventilatory support and survival at 28 days.

Investigators will also measure the proportion of patients experiencing significant asynchrony during the transition to spontaneous mechanical ventilation, who revert to sedation and controlled mechanical ventilation within the first 24 hours or at any point during mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with hypoxemic ARF, defined as a PaO2/FIO2 ratio <300 mmHg, under controlled invasive mechanical ventilation, with an expected duration of MV of at least 24h.
* Patients transitioning to spontaneous ventilation modes (PSV, PAV Plus, NAVA or APRV)

Exclusion Criteria:

* Tracheostomized patients.
* Decision not to maintain or add life support measures on the day of assessment (palliative care).
* Patient in ECMO.
* Air fistula or barotrauma that prevents adequate tidal volume monitoring.
* Severe injuries to the central nervous system that result in abolished or very high respiratory drive, for whom it is not possible to maintain protective tidal volume.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypoxemic ARF, defined as a PaO2/FIO2 ratio <300 mmHg, under controlled invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 422 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-06-12 (Estimated); Study Completion 2024-10-12 (Estimated)

PRIMARY OUTCOMES:
Low tidal volume | 24 hours
  Low tidal volume, defined as less or equal to 8 mLs per Kg of predicted body weight
Ventilator- free days | 28 days
  number of days alive and not receiving invasive mechanical ventilation after transition to spontaneous ventilation

SECONDARY OUTCOMES:
Hospital mortality | 28 days
  mortality in the hospital
Rate of patient-ventilator asynchrony | 24 hours
  presence of patient asynchrony 24h after transition to a spontaneous mode of mechanical ventilation
Number of participants that return to controlled mechanical ventilation in the first 24 hours | 24 hours
  return to controlled mechanical ventilation in the first 24 hours after transition to spontaneous ventilation
Number of participants that return to sedation in the first 24 hours | 24 hours
  return to sedation in the first 24 hours after transition to spontaneous ventilation
Number of participants that return to controlled mechanical ventilation after transition to spontaneous ventilation | 28 days
  return to controlled mechanical ventilation any time after transition to spontaneous ventilation
Number of participants that return to sedation after transition to spontaneous ventilation | 28 days
  return to sedation any time after transition to spontaneous ventilation
Number of participants with PEEP and FIO2 compatible with the ARDSnet PEEP/FIO2 table | 24 hours
  adherence to ARDSnet low PEEP/FIO2 table after transition to spontaneous ventilation
Number of participants who were extubated | 28 days
  Extubation and discontinuation of mechanical ventilation after the transition to spontaneous mode
Rate of reintubation | 28 days
  Reintubation after transition to spontaneous mode and extubation

CONTACTS AND LOCATIONS:
Overall Officials: JULIANA C FERREIRA, MD, Principal Investigator — University of Sao Paulo
Locations (10):
- Sanatorio Juncal SA, Buenos Aires, Argentina
- Hospital Municipal Boliviano Holandés, Universidad Mayor de San Andrés, La Paz, Bolivia
- Hospital das Clínicas -HCFMUSP, São Paulo, São Paulo, Brazil
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Clinica Universidad de la Sabana, Chía, Colombia
- Hospital Eugenio Espejo, Quito, Ecuador
- Hospital Civil Fray Antonio Alcalde, Guadalajara, Mexico
- Hospital San Roque, Asunción, Paraguay
- Hospital Rebagliati, Lima, Peru
- Hospital Espanol, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Undecided
data sharing will follow Institutional rules for patient data protection